CLINICAL TRIAL: NCT00594659
Title: Development and Efficacy Test of Computerized Treatment for Marijuana Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 88268; 1R01DA023526-01 (NIH); 1R01DA023526-02 (NIH); 1R01DA023526-03 (NIH)
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Results first posted 2013-12-04 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Marijuana Abuse and Dependence
Keywords: Marijuana; Treatment; Behavioral; Computer; Internet
MeSH Terms: conditions — Marijuana Abuse; Behavior | interventions — Psychotherapy; Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Therapist delivered cognitive behavioral treatment
  Interventions: Behavioral: Psychotherapy
- 2 (Experimental): Computerized Cognitive Behavioral treatment
  Interventions: Behavioral: Computerized Psychotherapy
- 3 (Active Comparator): Motivational enhancement therapy
  Interventions: Behavioral: Motivational enhancement therapy

INTERVENTIONS:
Behavioral: Psychotherapy — Nine session treatment
  Arms: 1
Behavioral: Computerized Psychotherapy — Nine session computer delivered treatment
  Arms: 2
Behavioral: Motivational enhancement therapy — Two session treatment
  Arms: 3

SUMMARY:
More US residents are dependent on marijuana than on any other illicit drug, and the number enrolled in treatment for marijuana continues to increase such that it is now comparable to that for cocaine and heroin. This application seeks to advance the overarching goal to develop and disseminate cost-effective treatments for marijuana dependence that can address this growing problem.

The researchers' previous research suggests that an intervention comprising motivational enhancement, cognitive-behavioral, and contingency-management components (MET/CBT/CM) produces greater rates of successful and durable outcomes than has been demonstrated previously. However, three issues relevant to its efficacy and eventual dissemination must be confronted. First, the outcomes achieved can only be characterized as modest; many individuals do not respond to the treatment and relapse rates remain problematic. Second, access is limited by the availability of trained providers. Third, the cost of delivering the treatment is higher than more traditional outpatient interventions.

To address these issues, Specific Aim 1 is to develop and test a computer-assisted version of MET/CBT/CM. Computerized treatments have the potential to increase overall effectiveness of treatment services by increasing availability of and access to potent treatments, and by applying innovative technology to enhance outcomes. During Year 1, the intervention will be developed and pilot tested. An interactive program that showed promise in a previous trial for opioid dependence will be modified and enhanced to deliver individualized MET/CBT/CM using effective computer learning technologies. These technologies and access to the MET/CBT/CM program made available via the Internet between treatment sessions and after treatment ends have the potential to promote better learning and more use of coping skills, which in turn can improve outcomes. During Years 2-4 a randomized trial will provide an initial efficacy test of cMET/CBT/CM by comparing it with a brief treatment (MET) and with therapist-delivered MET/CBT/CM. Specific Aim 2 is to learn more about how behavioral treatments like MET/CBT/CM work by focusing on two putative mechanisms of action examined in prior trials: self-efficacy/coping skills and impulsivity/delay discounting. The experimental design will provide a unique opportunity to explore such mechanisms in a novel context- where the therapist is vs. is not a prominent part of the treatment.

The proposed project will address the objectives of NIDA's Behavioral and Integrative Treatment Development Program by providing research on technology-assisted treatment that attempts to make treatment delivery less complex, easier to access, and less costly - while retaining or improving its effectiveness. Findings will inform future studies designed to refine the technology and how it is applied; conduct more definitive effectiveness testing; test generality to other populations including adolescents; and to further advance translation to community settings.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Meet criteria for current DSM-IV diagnosis of marijuana abuse or dependence
* Report use of marijuana on at least 40 of the past 90 days
* Severe psychological distress

Exclusion Criteria:

* Current dependence on alcohol or any other drug (except nicotine)
* Participation in treatment for alcohol/drug problem
* A legal status which will interfere with participation
* Plans to move out of the area in the next 12 months
* Living with someone who is already enrolled in the project
* Not living within approximately 30 miles of the research site
* Not being fluent in English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan J Budney, Ph.D., Principal Investigator — Dartmouth College
Locations (1):
- Geisel School of Medicine at Dartmouth, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment opened in November 2008 and closed in May 2011. Recruitment practices included newspaper and radio advertisements, flyers, and posters distributed in local businesses and agencies. The study took place at an outpatient psychiatry clinic.
Pre-assignment Details: Participants were excluded from trial prior to group assignment for at least one of the following:no evidence of marijuana use in at least 40 of the past 90 days prior to enrollment,participant met criteria for dependence on alcohol or illicit drugs,evidence of illicit drug use or K-2 use,interfering medical/psychiatric illness,or active refusal.
Groups:
- 1-MET/CBT/CM: Therapist delivered motivational enhancement therapy plus cognitive behavioral therapy plus contingency management (tMET/CBT/CM)
  Psychotherapy : Nine session treatment (wks 1-8 and wk 12)
  2x/wk urine drug testing
  Contingency Management voucher program
- 2-cMET/CBT/CM: Computer-delievered (c) MET/CBT/CM treatment
  Computerized Psychotherapy : Nine session computer delivered treatment
  2 times per week urine drug testing
- 3-tMET: Motivational enhancement therapy
  Motivational enhancement therapy : Two session treatment
  2x/wk urine drug testing
  non-contingent vouchers
Period: Overall Study
Arm/Group | 1-MET/CBT/CM | 2-cMET/CBT/CM | 3-tMET
Started | 29 | 30 | 16
Completed | 16 | 21 | 9
Not Completed | 13 | 9 | 7
Not completed — Lost to Follow-up | 13 | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- 1-MET/CBT/CM: Therapist delivered motivational enhancement therapy plus cognitive behavioral therapy plus contingency management (tMET/CBT/CM)
  Nine weekly therapy sessions delivered in weeks 1-8 and week 12
  2 times per week urine drug testing
  Contingency management program delivered monetary-based incentives contingent on each marijuana-negative urine toxicology test.
- 2-cMET/CBT/CM: Computer-delievered (c) MET/CBT/CM treatment
  Computer delivered nine MET/CBT sessions during weeks 1-8 and week 12. therapist delivered 3 brief supportive counseling sessions during weeks 1, 4, and 12.
  2 times per week urine drug testing.
  Contingency management program delivered monetary-based incentives contingent on each marijuana-negative urine toxicology test.
- 3-tMET: Therapist delivered motivational enhancement therapy (tMET)
  Two session treatment with sessions delivered during weeks 1 and 4.
  Two times per week urine drug testing.
  Non-contingent incentives delivered for attending each urine testing appointment.
- Total: Total of all reporting groups
Arm/Group | 1-MET/CBT/CM | 2-cMET/CBT/CM | 3-tMET | Total
Number analyzed (Participants) | 29 | 30 | 16 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 30 | 16 | 75
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (11.06) | 34.87 (11.07) | 35 (8.95) | 34.85 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 7 | 33
  Male | 17 | 16 | 9 | 42
Region of Enrollment [Number; unit: participants]
  United States | 29 | 30 | 16 | 75
Point prevalence abstinence [Number; unit: percentage of participants] — Total percentage column is not accurate because it is automatically summed, which results in an invalid number.
  percentage of participants | 0 | 13 | 12.5 | 25.5

OUTCOME MEASURES:

1. Primary Outcome: Consecutive Weeks of Marijuana Abstinence
Description: Longest period of marijuana abstinence achieved during the 12-week treatment period documented by urine testing and self-report.
Time Frame: From the start of treatment through the end of the active treatment period, i.e., 12 weeks.
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: consecutive weeks of abstinence
Groups:
- 1-tMET/CBT/CM: Therapist delivered cognitive behavioral treatment
  Psychotherapy : Nine session treatment
- 2-cMET/CBT/CM: Computerized Cognitive Behavioral treatment
  Computerized Psychotherapy : Nine session computer delivered treatment
- 3-tMET: Motivational enhancement therapy
  Motivational enhancement therapy : Two session treatment
Arm/Group | 1-tMET/CBT/CM | 2-cMET/CBT/CM | 3-tMET
Number analyzed (Participants) | 29 | 30 | 16
consecutive weeks of abstinence | 3.55 (4.39) | 2.82 (4.21) | 0.78 (1.97)
Statistical Analysis 1: Comparison: 1-tMET/CBT/CM vs 3-tMET; Pairwise comparison; non-parametric tests performed because of non-normal distribution; Test type: Superiority or Other; p < 0.05, accelerated bootstrapping
Statistical Analysis 2: Comparison: 2-cMET/CBT/CM vs 3-tMET; pairwise comparison; non-parametric analysis; Test type: Superiority or Other; p < .05, accelerated bootstrapping
Statistical Analysis 3: Comparison: 1-tMET/CBT/CM vs 2-cMET/CBT/CM; nonparametric pairwise comparison; non-normal distribution; Test type: Superiority or Other; p > 0.05, accelerated bootstrapping

2. Primary Outcome: Point Prevalence Abstinence Post Treatment
Description: Percent of participants that were marijuana abstinent based on urine toxicology testing at each follow up assessment across 9 month follow up period ( at the end of treatment, at 3-months, 6-months, and 9 months post the end of treatment).
Time Frame: 9 months (from the end of treatment to 9 months post-treatment).
Population: Intent to Treat
Measure: Number; unit: pecentage of participants abstinent
Arm/Group | 1-tMET/CBT/CM | 2-cMET/CBT/CM | 3-tMET
Number analyzed (Participants) | 29 | 30 | 16
pecentage of participants abstinent
  End of Treatment (ETX) Abstinence Rate | 44.8 | 46.7 | 12.5
  3-Months Post Treatment Abstinence Rate | 20.7 | 36.7 | 6.3
  6-months Post Treatment Abstinence Rate | 17.2 | 36.7 | 6.3
  9-months Post Treatment Abstinence Rate | 10.3 | 23.3 | 6.3
Statistical Analysis 1: Comparison: 1-tMET/CBT/CM vs 2-cMET/CBT/CM vs 3-tMET; pairwise comparisons among groups across 4 follow-up timepoints; Test type: Superiority or Other; p < 0.05, piecewise mixed model with logit link an; Performed across all assessments; Slope = 3.11, Standard Error of Mean 0.69 — Slope and p-value above are for group 1: baseline to ETX. Group 3 vs. Group 1 baseline to ETX slope, p < 0.05. All other pairwise comparisons p > 0.05

ADVERSE EVENTS:
Arm/Group | 1-MET/CBT/CM | 2-cMET/CBT/CM | 3-tMET
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30 | 0/16
Other Adverse Events (participants affected / at risk) | 0/29 | 0/30 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No